CLINICAL TRIAL: NCT00415025
Title: Evaluation of Normal Tissue Toxicities in Head and Neck Cancer Patients Receiving Intensity Modulated Radiotherapy (IMRT)
Brief Title: Side Effects of High-Dose Intensity-Modulated Radiation Therapy in Treating Patients With Advanced Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: H-2004-0168; P30CA014520 (NIH); WCCC-RO-03313; CDR0000515323; NCT00214188 (obsolete NCT alias)
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Head and Neck Cancer; Long-term Effects Secondary to Cancer Therapy in Adults; Oral Complications of Radiation Therapy; Radiation Toxicity
Keywords: long-term effects secondary to cancer therapy in adults; oral complications of radiation therapy; radiation toxicity; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III basal cell carcinoma of the lip; stage III squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV squamous cell carcinoma of the lip and oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; recurrent lymphoepithelioma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — Chemotherapy, Adjuvant; Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Procedure: adjuvant therapy
Procedure: management of therapy complications
Procedure: quality-of-life assessment
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Tests that measure how much saliva is made, hearing, swallowing, voice function, and quality of life may improve the ability to plan treatment for patients with advanced head and neck cancer and may help doctors find better ways to treat the cancer.

PURPOSE: This clinical trial is studying the side effects of high-dose intensity-modulated radiation therapy in treating patients with advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess salivary function in patients with advanced head and neck cancer treated with intensity-modulated radiotherapy (IMRT) by measuring stimulated saliva production at 6 and 12 months after completion of therapy.
* Compare salivary function in these patients to salivary function in historical controls.

Secondary

* Assess auditory, swallow, and voice function and quality of life of these patients before and after IMRT or chemoradiotherapy.
* Advance experience with IMRT/tomotherapy and improve field design for irradiating head and neck cancer in an effort to reduce radiation dose and minimize effects on surrounding normal tissue.

OUTLINE: This is a prospective study.

Patients undergo standard of care high-dose intensity-modulated radiotherapy (IMRT) to the head and neck.

Patients undergo baseline and post-treatment testing of auditory, salivary, swallow, and voice function as well as quality of life evaluation.

Patients are evaluated for radiation-induced toxicities at 1, 6, and 12 months after completion of IMRT.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced head and neck cancer
* Indication for radiotherapy or chemoradiotherapy as primary or postoperative therapy AND meets 1 of the following criteria:

  * More than 75% of bilateral parotid glands expected to receive ≥ 45 cGy of radiation using conventional treatment field design
  * Either or both central auditory apparatus predicted to receive > 45 cGy of radiation

PATIENT CHARACTERISTICS:

* No comorbid medical condition that would preclude radiotherapy
* No serious concurrent psychosocial, familial, sociological, geographical, or other condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-06; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Stimulated saliva production at 6 months after completion of intensity-modulated radiotherapy (IMRT)
Comparison of salivary function of patients in current study to salivary function of historical controls

SECONDARY OUTCOMES:
Auditory, swallow, and voice function at 6 months after completion of IMRT
Quality of Life (QOL) as assessed at baseline and at 1, 6, and 12 months after completion of IMRT
Toxicities as measured by NCI CTCAE v3.0
Improvement in IMRT/tomotherapy field design

CONTACTS AND LOCATIONS:
Overall Officials: Paul M. Harari, MD, Study Chair — University of Wisconsin, Madison